CLINICAL TRIAL: NCT06377176
Title: Massage Therapy for Infants and Mothers
Brief Title: Postpartum Massage Therapy for Women and Infants: The Effect on Maternal Depression, Stress, Fatigue and Infant Temperament
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Principal Investigator, Evi Nurhidayati, Principal Investigator, National Taipei University of Nursing and Health Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NTUNHSEN
Record Dates: First submitted 2024-03-04; First posted 2024-04-22 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Postpartum Depression
Keywords: Massage Therapy; Postpartum Depression; Stress; Fatigue; Infant Temperament
MeSH Terms: conditions — Depression, Postpartum; Fatigue | interventions — Massage

STUDY DESIGN:
Intervention Model Description: A quasi-experimental design was utilized in this investigation; it comprised a pre-test and a post-test administered to two distinct groups. The intervention group was subjected to pre-testing before receiving the intervention, and after the intervention, mother and infant massage treatment was delivered to the intervention group. Post-testing was performed on both groups, with the control group receiving mother and infant massage.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Massage therapy for mother and infant.
  Interventions: Other: Massage therapy
- Control group (No Intervention): the control group received standard care.

INTERVENTIONS:
Other: Massage therapy — the intervention group underwent ten sessions of twice-weekly mother and infant massage therapy for five weeks.
  Arms: Intervention group

SUMMARY:
Mother and infant massage, a type of complementary therapy, possesses the capacity to ameliorate maternal depression, stress, fatigue, and also infant temperaments and convert them into more manageable ones. The objective of this study was to determine the effect of mother and infant massage therapy on maternal depression, stress, fatigue, and infant temperament. In this quasi-experimental study, a total of 102 participants were allocated into two groups based on a pretest and posttest. During a period of five weeks, the experimental groups were subjected to ten massages per week, twice every week. On the data, a generalized estimating equation (GEE) was implemented. This study's hypothesis was an improvement in maternal depression, stress, fatigue, and infant temperament.

DETAILED DESCRIPTION:
Data collection procedures Preparation stage Two research assistants with a master's degree in midwifery and two years of clinical experience were chosen by the researcher. The researcher describes and discusses the purpose, intervention protocol, research instrument, and COVID-19 protocol of the study. All research assistants as data collectors and the therapist are required to have received either two doses of the COVID-19 vaccine or a handwash or hand sanitizer, in addition to wearing a face mask. Furthermore, the research assistant requested to accompany the researcher as they conducted the informed consent and questionnaire administration process with the participant on an estimated three separate occasions. The research assistant conducted an informed consent test on the participants after three observations; individuals who adequately showcased their ability were granted employment as research assistants. Daily activity logs must be included on self-report forms completed by the research assistant.

Additionally, the researcher designates the mother and infant massage therapist; for the baby massage, the researcher collaborates with a physiotherapist and midwives who possess more than two years of clinical experience and a midwife who holds certification in baby massage therapy. Following this, the massage therapist and researcher demonstrated and discussed the massage technique with the mother and child. During the intervention, the researcher additionally provided the mothers with a baby doll so that they could serve as models for baby massage to the mothers while the physiotherapists or midwives attended to the infants. Upon the conclusion of the intervention, the mothers would be capable of performing massage independently.

Implementation stage The researcher employed the EPDS questionnaire as a screening tool to identify postpartum mothers for depression; participants were chosen based on their EPDS score of 13. Following this, the investigator proceeds to deliver an elucidation of the study's aims and methodology to the participant. On the day of the questionnaire's initiation, the consent form is duly signed by the respondent. The research assistant confirmed the questionnaire's completion upon its return and requested that the respondents complete it, including the respondent code, and place it in the file holder.

Following the completion of the initial questionnaires by both groups during the meeting, the intervention group underwent ten sessions of twice-weekly mother and infant massage therapy over the course of five weeks. The mother promptly resubmits the questionnaires following the conclusion of the newborn massage therapy. A month later, the mother proceeds to complete the remaining questionnaires.

A regimen for the respondent and therapist to receive massages was formulated by the researcher. The receiver dictates the duration of the massage. The researcher then created a massage regimen to be executed twice weekly for five weeks. Respondents 1 through 30 adhered to a Monday through Thursday routine, but those 31 through 52 observed Tuesday through Friday. Four to six participants were massaged per therapist, and a total of seven therapists were hired. The massage hours of operation are from 7:00 am to 5:00 pm. A two-hour period separated each responder; for instance, in the scenario where one respondent received a massage at 7:00 am, the subsequent respondent would receive one at 9:00 am.

The control group is administered standard care or routine mother and infant care. As part of usual care, the CHC midwife conducts routine assessments of the infant's height and weight, in addition to furnishing the mother with relevant information. Furthermore, after completing the second posttest, mother and infant massage therapy is implemented for the control group.

Sample size This research uses G-power calculation to examine the number of samples needed. Based on the G-power calculation and the assumption of a minimum medium effect size of 0.25% at a significance level of 0.05 and 80% power, an estimated sample size of 86 participants is necessary. Considering a 20 percent attrition rate, 104 individuals were recruited in total. By utilizing convenience sampling, this research incorporates all eligible participants. Two participants were ineligible to participate in this research due to a family-related concern.

Data analysis The data was analyzed by univariate, bivariate, and multivariate. Bivariate statistics using independent t-tests, Chi-square, Fisher exact test, Pearson correlation; and for the multivariate data using generalized estimated equation.

ELIGIBILITY:
Inclusion Criteria:

* Edinburgh Postnatal Depression Scale (EPDS) score more and equal to 13.
* Must be able to read.
* All types of delivery.
* Full-term gestation.
* Healthy infant.

Exclusion Criteria:

* Drug abuse history.
* Bipolar.
* Schizophrenia history.

Ages: 1 Month to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 102 (Actual)
Dates: Start 2021-06-16 (Actual); Primary Completion 2021-10-03 (Actual); Study Completion 2021-10-03 (Actual)

PRIMARY OUTCOMES:
Depression | Pretest: At the initial encounter, eligible as a respondent and agreed to participate in the research then fill out the questionnaires. Posttest 1: after the end of massage therapy session (5 weeks). Posttest 2: 1 month after posttest 1.
  Score of mother depression on postpartum. EPDS score greater than or equal to 13.

SECONDARY OUTCOMES:
Stress | Pretest: At the initial encounter, eligible as a respondent and agreed to participate in the research then fill out the questionnaires.. Posttest 1: after the end of massage therapy session (5 weeks). Posttest 2: 1 month after posttest 1.
  The score of mother's stress. PSS-14 score range from 0-56. High scores indicate more stress.
Fatigue | Pretest: At the initial encounter, eligible as a respondent and agreed to participate in the research then fill out the questionnaires.. Posttest 1: after the end of massage therapy session (5 weeks). Posttest 2: 1 month after posttest 1.
  The score of mothers fatigue. Fatigue scores range from 0-10. High Scores indicate more fatigue.
Infant temperament | Pretest: At the initial encounter, eligible as a respondent and agreed to participate in the research then fill out the questionnaires.. Posttest 1: after the end of massage therapy session (5 weeks). Posttest 2: 1 month after posttest 1.
  The score of infant temperament. Infant temperament score 0-3. High scores indicate as a difficult temperament.

CONTACTS AND LOCATIONS:
Locations (1):
- Community Health Center, Sleman, Special Region of Yogyakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No